CLINICAL TRIAL: NCT02037633
Title: Fascia Iliaca Compartment Block Versus Fentanyl for Positioning Patients With Hip Fractures for Central Nervous Blockade: a Randomized Trial.
Brief Title: Analgesia for Positioning Hip Fracture Patients for Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Maria Diakomi, MD, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 478-9227/25-7-2012
Record Dates: First submitted 2014-01-12; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Fentanyl; Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fascia iliaca compartment block (Active Comparator)
  Interventions: Procedure: Fascia iliaca compartment block; Drug: ropivacaine
- Fentanyl (Active Comparator)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl IV
  Arms: Fentanyl
Procedure: Fascia iliaca compartment block — Fascia iliaca compartment block using ropivacaine
  Arms: Fascia iliaca compartment block
Drug: ropivacaine
  Arms: Fascia iliaca compartment block

SUMMARY:
The purpose of this study is to compare two analgesic methods performed preoperatively to assist positioning patients for performance of spinal anesthesia, namely fascia iliaca blockade and intravenous fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture

Exclusion Criteria:

* contraindications for central nervous blockade
* impaired cognition or dementia
* multiple fractures
* any previous analgesic administration during the last 12 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pain scores on the Numeric Rating Scale | Group A: 5 minutes after intervention (fentanyl), Group B: 20 minutes after intervention (block)

SECONDARY OUTCOMES:
Duration of spinal anesthesia performance | Group A: 5 minutes after intervention (fentanyl), Group B: 20 minutes after intervention (block)
  It will be measured in "minutes", from the start of positioning maneuvers to the spinal needle removal
Quality of patient's position | Group A: 5 minutes after intervention (fentanyl), Group B: 20 minutes after intervention (block)
  The position will be characterized as "unsatisfactory", "satisfactory", "good" or "very good"

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepieion Hospital of Voula, Athens, Attica, Greece

REFERENCES:
- [Background] Yun MJ, Kim YH, Han MK, Kim JH, Hwang JW, Do SH. Analgesia before a spinal block for femoral neck fracture: fascia iliaca compartment block. Acta Anaesthesiol Scand. 2009 Nov;53(10):1282-7. doi: 10.1111/j.1399-6576.2009.02052.x. Epub 2009 Jul 22. PMID 19650803
- [Background] Hogh A, Dremstrup L, Jensen SS, Lindholt J. Fascia iliaca compartment block performed by junior registrars as a supplement to pre-operative analgesia for patients with hip fracture. Strategies Trauma Limb Reconstr. 2008 Sep;3(2):65-70. doi: 10.1007/s11751-008-0037-9. Epub 2008 Sep 2. PMID 18762870
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043